CLINICAL TRIAL: NCT01510704
Title: Randomised, Double-blind, Placebo-controlled, Dose-ranging Phase II Study of APD421 for the Prevention of Post-operative Nausea and Vomiting
Brief Title: Phase II Dose-ranging Study of APD421 in PONV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DP10006
Record Dates: First submitted 2012-01-12; First posted 2012-01-16 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Low dose APD421 (Experimental): 1mg dose level
  Interventions: Drug: APD421
- Mid Dose APD421 (Experimental): 5mg dose level
  Interventions: Drug: APD421
- High Dose APD421 (Experimental): 20mg dose level
  Interventions: Drug: APD421

INTERVENTIONS:
Drug: APD421 — IV
  Arms: High Dose APD421; Low dose APD421; Mid Dose APD421
Drug: Placebo — IV
  Arms: Placebo

SUMMARY:
To assess the efficacy and safety of different doses of APD421 in the prevention of post-operative nausea and vomiting (PONV) in adult patients at moderate to high-risk of PONV. Patients must be undergoing elective surgery under general anaesthesia (hysterectomy (any surgical technique), cholecystectomy (any surgical technique) or "other" elective surgery scheduled to last at least one hour from induction of anaesthesia), requiring at least one overnight stay in hospital, and have at least 2 of the following risk factors for PONV: Past history of PONV and/or motion sickness; Non-smoking status; Female gender; Planned opiate use for post-operative analgesia.

ELIGIBILITY:
Inclusion criteria

1. Male or female patients ≥ 18 years of age
2. Ability and willingness to give written informed consent
3. Patients undergoing elective surgery under general anaesthesia requiring at least one overnight stay in hospital for either:

   1. Hysterectomy (any surgical technique)
   2. Cholecystectomy (any surgical technique)
   3. Other elective surgery requiring overnight admission to hospital and scheduled to last at least 1 hour from induction of anaesthesia
4. Patients with at least 2 of the following risk factors for PONV:

   1. Past history of PONV and/or motion sickness
   2. Habitual non-smoking status
   3. Female sex
   4. Expected to receive opioid analgesia post-operatively
5. American Society of Anesthesiologists (ASA) risk score I-III
6. Adequate cardiac, hepatic and renal function

   * QTc interval < 500 ms
   * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) < 5 x upper limit normal (ULN)
   * Bilirubin < 3 x ULN
   * Creatinine < 2 x ULN
7. Adequate haematological function

   * Haemoglobin ≥ 9 g/dL
   * White blood count ≥ 3.0 x 109/L
   * Platelet count ≥ 100 x 109/L
8. For females of child-bearing potential: ability and willingness to use a highly effective form of contraception (e.g., abstinence from sexual intercourse, surgical sterilisation (of subject or partner) or a double-barrier method of contraception such as either an intra-uterine device (IUD) or an occlusive cap with spermicide, in conjunction with partner's use of a condom) between the date of screening and at least 48 hours after administration of study drug.

Exclusion Criteria

1. Patients undergoing outpatient/day case surgery
2. Patients undergoing surgery where the patient is expected to remain ventilated for a period after surgery
3. Patients undergoing intra-thoracic, transplant or central nervous system surgery
4. Patients receiving a local anaesthetic/regional neuraxial (intrathecal or epidural) block
5. Patients who are expected to need a naso- or oral-gastric tube in situ after surgery is completed
6. Patients receiving the active ingredient of APD421 for any indication within the last 2 weeks
7. Patients who are allergic to the active ingredient or any of the excipients of APD421
8. Patients with a pre-existing vestibular disorder or history of dizziness
9. Patients with pre-existing nausea or vomiting in the 24 hours before surgery
10. Patients treated with regular anti-emetic therapy including corticosteroids
11. Patients being treated with medications which could induce torsades de pointes, including Class Ia antiarrhythmic agents such as quinidine, disopyramide, procainamide; Class III antiarrhythmic agents such as amiodarone and sotalol; and other medications such as bepridil, cisapride, thioridazine, methadone, IV erythromycin, IV vincamine, halofantrine, pentamidine, sparfloxacin
12. Patients being treated with levodopa
13. Patients who are pregnant or breast feeding
14. Patients with a history of alcohol abuse
15. Patients with pre-existing, clinically significant cardiac arrhythmia
16. Patients diagnosed with Parkinson's disease
17. Patients who have received anti-cancer chemotherapy in the previous 4 weeks
18. Patients with a history of epilepsy
19. Any other concurrent disease or illness that, in the opinion of the investigator makes the patient unsuitable for the study
20. Patients who have participated in a previous study within the last 28 days (French sites only: Patients who have participated in a previous study within the last 6 months, if required by national or local regulations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kranke, MD, Principal Investigator — University Hospitals of Würzburg
Locations (13):
- Duke University Medical Center, Durham, North Carolina, United States
- France (6):
  - University Hospital, Besançon
  - Hôpital mère enfant, Bron
  - Hôpital Huriez, Lille
  - University Hospital, Nancy
  - Hôpital FOCH, Paris
  - Hautepierre Hospital, Strasbourg
- Germany (6):
  - HELIOS Klinikum Aue, Aue
  - Charité - Universitätsmedizin, Berlin
  - Universität Heidelberg, Heidelberg
  - Klinikum Ludwigshafen, Ludwigshafen
  - Philipps University, Marburg
  - University Hospitals of Würzburg, Würzburg

REFERENCES:
- [Derived] Kranke P, Eberhart L, Motsch J, Chassard D, Wallenborn J, Diemunsch P, Liu N, Keh D, Bouaziz H, Bergis M, Fox G, Gan TJ. I.V. APD421 (amisulpride) prevents postoperative nausea and vomiting: a randomized, double-blind, placebo-controlled, multicentre trial. Br J Anaesth. 2013 Dec;111(6):938-45. doi: 10.1093/bja/aet251. Epub 2013 Jul 19. PMID 23872464

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Single-dose IV placebo
- Low Dose APD421: Single-dose 1 mg IV APD421
- Mid Dose APD421: Single-dose 5 mg IV APD421
- High Dose APD421: Single-dose 20 mg IV APD421
Period: Overall Study
Arm/Group | Placebo | Low Dose APD421 | Mid Dose APD421 | High Dose APD421
Started | 54 | 58 | 50 | 53
Completed | 54 | 58 | 50 | 53
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose APD421 | Mid Dose APD421 | High Dose APD421 | Total
Number analyzed (Participants) | 54 | 58 | 50 | 53 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (13.6) | 50 (14.5) | 50 (16.2) | 50.7 (15.7) | 49.9 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 53 | 48 | 49 | 197
  Male | 7 | 5 | 2 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Nausea or Vomiting
Time Frame: 24 hours
Population: ITT
Measure: Number; unit: participants
Arm/Group | Placebo | Low Dose APD421 | Mid Dose APD421 | High Dose APD421
Number analyzed (Participants) | 54 | 58 | 50 | 53
participants | 37 | 28 | 20 | 30

ADVERSE EVENTS:
Arm/Group | Placebo | Low Dose APD421 | Mid Dose APD421 | High Dose APD421
Serious Adverse Events (participants affected / at risk) | 2/54 | 1/58 | 0/50 | 2/53
Other Adverse Events (participants affected / at risk) | 52/54 | 50/58 | 39/50 | 46/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | Low Dose APD421 (N=58) | Mid Dose APD421 (N=50) | High Dose APD421 (N=53)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WOUND HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=54) | Low Dose APD421 (N=58) | Mid Dose APD421 (N=50) | High Dose APD421 (N=53)
Procedural Pain (Injury, poisoning and procedural complications) | 28 (28) | 30 (30) | 27 (27) | 27 (27)
Nausea (Gastrointestinal disorders) | 28 (28) | 19 (19) | 13 (13) | 24 (24)
Vomiting (Gastrointestinal disorders) | 18 (18) | 14 (14) | 7 (7) | 9 (9)
Constipation (Gastrointestinal disorders) | 6 (6) | 6 (6) | 6 (6) | 6 (6)
Flatulence (Gastrointestinal disorders) | 7 (7) | 7 (7) | 4 (4) | 4 (4)
Pain (General disorders) | 5 (5) | 7 (7) | 3 (3) | 6 (6)
Procedural nausea (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | 4 (4) | 5 (5)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No